CLINICAL TRIAL: NCT00319137
Title: A Randomized, Single-Blind, Single-Attack, Placebo-Controlled, Adaptive Design Study to Assess the Safety and Efficacy of Doses of 5-180 mg of the iNOS Inhibitor GW274150 in the Treatment of Acute Migraine During the Mild Headache Phase
Brief Title: An Adaptive Design Trial Of GW274150 In The Treatment Of Acute Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NOS102512
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Migraine Disorders; Migraine
Keywords: GW274150; Nitric Oxide; acute migraine
MeSH Terms: conditions — Migraine Disorders | interventions — GW 274150

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW274150

SUMMARY:
Nitric oxide (NO) is likely to be involved in the development of migraine headache. Nitric oxide synthase (NOS) is an important chemical involved in the production of NO. Reduction of NOS, and therefore NO, may be an effective technique for the treatment of migraine headache. GW274150 is a highly selective inhibitor of NOS and offers the potential of anti-inflammatory activity in migraine through a novel mechanism of action. The intent of this study is to investigate the safety and efficacy of GW274150 for the acute treatment of migraine headache.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from migraine with or without aura.
* Migraine for at least one year, and the age of onset was prior to 50 years.
* Consistent migraine headache over time and has had at least 1 migraine headache attacks but less than 15 days with headache (migraine or non-migraine) per month in each of the three months prior to the Screening Visit and maintains this requirement during the baseline period.
* Able to distinguish migraine headache attacks as discreet attacks from other headaches (i.e. tension-type headaches).
* Typically have moderate to severe migraine pain preceded by an identifiable mild pain phase.
* No clinically significant abnormality identified on the medical or laboratory evaluation. A subject with a clinical abnormality or laboratory parameters outside the reference range may be included only if the doctor considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* Written informed consent prior to entry into the study.
* Females who are: a) non-childbearing potential or, b) of child-bearing potential, has a negative pregnancy test at screen, and is taken adequate contraceptive measures.

Exclusion Criteria:

* As a result of the medical interview, physical examination or screening investigations, that the doctor considers the subject unfit for the study.
* History of alcohol, substance or drug abuse within the last year.
* Taken a migraine prophylactic medication within 1 month of the Screening Visit.
* Uses an opiate as first line acute treatment for migraine attacks.
* History of ergotamine, triptan, opioid, or combination medication intake on greater than/equal 10 days per month on a regular basis for greater than/equal 3 months.
* History of simple analgesic intake on greater than/equal 15 days per month for greater than/equal 3 months.
* Do not receive migraine relief from a triptan migraine treatment.
* Uncontrolled hypertension at the Screening Visit, defined as systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg.
* Evidence of renal impairment - calculated creatinine clearance <60ml/min or clinically relevant finding on urinalysis.
* History of drug or other allergy which, in the opinion of the doctor, makes the subject unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126
Dates: Start 2005-12

PRIMARY OUTCOMES:
Dose of GW274150 that results in 50% of subjects reporting cessation of migraine pain by 2 hours and to study the relationship between dose and therapeutic response.

SECONDARY OUTCOMES:
Adverse events following treatment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Adelaide, South Australia, Australia
- New Zealand (4):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Wellington